CLINICAL TRIAL: NCT05111145
Title: A Phase 3b Open-label Study Evaluating the Safety of Elexacaftor/Tezacaftor/Ivacaftor Combination Therapy in Subjects With Cystic Fibrosis
Brief Title: A Study Evaluating the Safety of Elexacaftor/Tezacaftor/Ivacaftor in Participants With Cystic Fibrosis (CF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX20-445-121; 2020-004885-21 (EudraCT Number)
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Results first posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-06

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — elexacaftor, ivacaftor, tezacaftor drug combination; ivacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ELX/TEZ/IVA (Experimental): Participants received ELX 200 mg once daily (qd)/TEZ 100 mg qd/IVA 150 mg every 12 hours (q12h) in the treatment period for up to 36 weeks.
  Interventions: Drug: ELX/TEZ/IVA; Drug: IVA

INTERVENTIONS:
Drug: ELX/TEZ/IVA — Fixed-dose combination tablets for oral administration.
  Other Names: VX-445/VX-661/VX-770; elexacaftor/tezacaftor/ivacaftor
Drug: IVA — Tablets for oral administration.
  Other Names: VX-770; ivacaftor

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of elexacaftor (ELX)/tezacaftor (TEZ)/ivacaftor (IVA) in participants with CF who are 12 years of age or older.

ELIGIBILITY:
Key Inclusion Criteria:

* Completed study drug treatment in parent study (VX19-445-117 [NCT04599465] or VX20-445-126 [NCT04969224]), or had study drug interruption(s) in parent study but completed study visits up to the last scheduled visit of the treatment period in the parent study

Key Exclusion Criteria:

* History of drug intolerance in a parent study

Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Australia (7):
  - The Prince Charles Hospital, Chermside
  - Alfred Hospital, Melbourne
  - Institute for Respiratory Health, Nedlands
  - Telethon Kids Institute, Nedlands
  - The Royal Children's Hospital, Parkville
  - Mater Adult Hospital, South Brisbane
  - Queensland Children's Hospital, South Brisbane
- Belgium (4):
  - Cliniques Universitaires de Bruxelles Hopital Erasme, Brussels
  - Universitair Ziekenhuis Brussel - Campus Jette, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Universitaire Ziekenhuizen Leuven - Campus Gasthuisberg, Leuven
- Canada (3):
  - University of Calgary Medical Clinic of the Foothills Medical Centre, Calgary
  - Stollery Children's Hospital, Edmonton
  - Queen Elizabeth II Health Sciences Center, Halifax
- Czechia (2):
  - Klinika Nemoci Plicnich a Tuberkulozy, Brno
  - Fakultni nemocnice v Motole, Prague
- Spain (8):
  - Hospital Saint Joan de Deu, Barcelona
  - Hospital Universitari Vall d Hebron, Barcelona
  - Hospital Universitari Vall d´Hebron Servicio de Broncoscopia, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Virgen de la Arrixaca, Murcia
  - Corporacio Sanitaria Parc Tauli - Sabadell Hospital Universitari, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants from Parent Studies VX19-445-117 (NCT04599465) and VX20-445-126 (NCT04969224) were enrolled in this study. A total of 86 participants were enrolled in this study.
Groups:
- ELX/TEZ/IVA: Participants received elexacaftor (ELX) 200 mg once daily (qd)/tezacaftor (TEZ) 100 mg qd/ivacaftor (IVA) 150 mg every 12 hours (q12h) in the treatment period for up to 36 weeks.
Period: Overall Study
Arm/Group | ELX/TEZ/IVA
Started | 86
Completed | 0
Not Completed | 86
Not completed — Commercial drug is available for participant | 76
Not completed — Participant enrolled in another qualified Vertex study | 10

BASELINE CHARACTERISTICS:
Population: Baseline data is based on the parent study baseline, which is defined as the most recent non-missing measurement collected before the first dose of study drug in the treatment period of parent studies. Baseline data is presented for participants who received at least 1 dose of study drug in this study
Groups:
- ELX/TEZ/IVA: Participants received ELX 200 mg qd/TEZ 100 mg qd/IVA 150 mg q12h in the treatment period for up to 36 weeks.
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 49
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 79
  Black or African American | 0
  Asian | 0
  American Indian or Alaska Native | 0
  Native Hawaiian or other Pacific Islander | 0
  Other | 0
  Not collected per local regulations | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 11
  Not Hispanic or Latino | 68
  Not collected per local regulations | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability as Assessed by Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Day 1 up to Week 36
Population: Safety set included for all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | ELX/TEZ/IVA
Number analyzed (Participants) | 86
Participants
  Participants with TEAEs | 61
  Participants with SAEs | 4

ADVERSE EVENTS:
Time Frame: Day 1 up to Week 36
Arm/Group | ELX/TEZ/IVA
All-Cause Mortality (participants affected / at risk) | 0/86
Serious Adverse Events (participants affected / at risk) | 4/86
Other Adverse Events (participants affected / at risk) | 33/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=86)
Gastroenteritis viral (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ELX/TEZ/IVA (N=86)
COVID-19 (Infections and infestations) | 16
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 11
Nasopharyngitis (Infections and infestations) | 9
Upper respiratory tract infection (Infections and infestations) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/45/NCT05111145/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-12): https://cdn.clinicaltrials.gov/large-docs/45/NCT05111145/SAP_001.pdf